CLINICAL TRIAL: NCT02730845
Title: Intra-articular Versus Intravenous Administration of Dexmedetomidine in Arthroscopic Knee Surgeries: A Prospective Randomized Study
Brief Title: Intra-articular Versus Intravenous Dexmedetomidine in Arthroscopic Knee Surgeries Under Local Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: R∕ 15.10.40
Record Dates: First submitted 2016-02-11; First posted 2016-04-07 (Estimated); Last update posted 2020-09-22 (Actual); Status verified 2020-09

CONDITIONS: Knee Arthroscopy
Keywords: Elective; local anesthesia; knee arthroscopy; Dexmedetomidine
MeSH Terms: interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intra-articular dexmedetomidine (Active Comparator): Patients will be subjected for elective knee arthroscopy under local anesthesia (Intra-articular dexmedetomidine + Intra-articular bupivacaine).
  Interventions: Drug: Intra-articular dexmedetomidine
- Intravenous dexmedetomidine (Placebo Comparator): patients will be subjected for elective knee arthroscopy under local anesthesia (i.v. dexmedetomidine + Intra-articular bupivacaine).
  Interventions: Drug: Intravenous dexmedetomidine

INTERVENTIONS:
Drug: Intra-articular dexmedetomidine — Patients will receive an intra-articular mixture of 19 ml bupivacaine 0.5% with epinephrine 1:200.000 added to 1ml (1 µg/kg) of dexmedetomidine (total volume 20 ml), and i.v. saline 20 ml infused over 10 min starting with local anesthesia
  Arms: Intra-articular dexmedetomidine
Drug: Intravenous dexmedetomidine — Patients will be injected intra-articularly with mixture of 19 ml 0.5% bupivacaine with epinephrine 1:200.000 and 1 ml of isotonic saline (total volume 20 ml), in addition to i.v. 20 ml saline containing 1 µg/kg dexmedetomidine over 10 min infusion starting with local anesthesia.
  Arms: Intravenous dexmedetomidine

SUMMARY:
The present study will be carried to evaluate the efficacy of intra-articular 0.5 bupivacaine with intra-articular or intravenous alpha-2agonist; Dexmedetomidine; for intraoperative anesthesia and postoperative analgesia after arthroscopic knee surgery.

Arthroscopic knee surgery is one of the most common minimally invasive orthopedic procedures in recent practice which is frequently performed as a day surgery procedures. It can be done under general, regional or local anesthesia (LA) with or without sedation. It is associated with varying amount of postoperative pain. Postoperative pain negatively influences patient's early ambulation, rehabilitation and psychology which consecutively prolonged the hospital stay.

Intra-articular administration of local anesthetic for knee arthroscopy is a well-documented procedure that offers many advantages over other anesthesia types. Many anesthesiologists are still trying to improve the technique of local anesthetic administration through using many combinations with LA solutions in order to administer safe anesthesia to those patients and to obtain a pain-free knee with good operating conditions.

Dexmedetomidine is a highly selective α2 adrenergic agonist. It has analgesic, sedative, anxiolytic, hypnotic, sympatholytic, antihypertensive properties with anesthetic sparing effects. It becomes an attractive alternative to the current opioids because it does not have a respiratory depressant or addictive effect.

DETAILED DESCRIPTION:
All patients were kept fasting after midnight and received midazolam 5 mg orally as premedication. All patients were premedicated with I.V. midazolam 0.03 mg/kg ten minutes before starting the operation. The anesthetic technique was standardized for all patients. All surgical procedures were performed by the same surgeon and consisted of arthroscopic removal of torn meniscus. Both intra-articular and intravenous solutions were prepared by an individual not involved in the study and the intra-articular drugs were injected by the surgeon (without knowing the contents). The anesthesiologist managing and monitoring the patient throughout the surgery provides IV drugs. No leg holder or tourniquet or surgical drain was used for any of the cases. After preparation and draping the patient's leg, patients were warned prior to each needle stick to decrease anxiety. All procedures were performed under complete aseptic conditions. Skin and subcutaneous tissues at each arthroscopic portal site were anesthetized with LA consisting of injection of a mixture of 2% lidocaine 5 mL with 1:200,000 epinephrine.

Care should be taken to avoid infiltration of the fat pad. It is a relatively aneural structure; as, too much local infiltration allows it to bulge out into the joint during the surgery. Flexion and extension of the knee joint several times help to spread of intra-articular solution and then waiting 20 minutes for anesthesia to take effect is helpful before the surgical incision.

The arthroscope was inserted into the knee, and inflow through the sheath was established. No pump was used for the saline inflow which was maintained through the arthroscope by the gravity. Gravity outflow drained through the superolateral portal. A separate egress cannula was used if indicated. The patient was encouraged to view the video monitor during the procedure. Constant verbal communication between the surgeon and the patient is important throughout the arthroscopic examination and surgery. This keeps the patient anxiety and muscle tension to the minimum which facilitates manipulation of the leg and thorough examination of the entire joint. Once finishing, instruments were removed and portals were closed with a 4-0 absorbable suture subcutaneously and steri-strips. A compression dressing was applied for three days to the knee.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists physical status I or II
* Patients scheduled for elective unilateral knee arthroscopy

Exclusion Criteria:

* Refusal of local anesthesia
* History of cardiovascular disease
* History of cerebrovascular disease
* History of respiratory diseases
* History of impaired renal functions
* History of impaired hepatic functions
* Pregnancy
* Allergy to the study drugs
* Uncontrolled diabetes
* Coagulopathies
* Hypertension treated with α methyldopa, clonidine or β adrenergic blockers
* Patients receiving chronic pain treatment
* Patients receiving psychoactive drugs
* Patients receiving anticoagulant drugs
* Prior ipsilateral knee surgery
* Infection at site of injection

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2015-12-01 (Actual); Primary Completion 2016-04-01 (Actual); Study Completion 2016-05-30 (Actual)

PRIMARY OUTCOMES:
Pain scores | for 24 hours starting immediately before performing the procedure
  Pain will be assessed using 10 cm visual analogue scale (VAS)

SECONDARY OUTCOMES:
Heart rate | starting immediately before performing the procedure
Blood pressure | starting immediately before performing the procedure
  Changes in systolic and mean blood pressure
Oxygen saturation | starting immediately before performing the procedure
  Changes in peripheral oxygen saturation
Respiratory rate | starting immediately before performing the procedure
  Changes in respiratory rates will be recorded
Level of sedation | For 24 hours after performing the injection
  will be evaluated using the following scale: (5= awake/alert to 0= asleep/unarousable )
Patient Satisfaction Score | For 24 hours after performing the procedure
  will be assessed using the following scale: 5= very satisfied, 4= satisfied, 3 = neutral, 2 = dissatisfied,
  1 = very dissatisfied
Time to first postoperative analgesic requirement | For 24 hours after performing the injection
  This will be recorded as the time to first postoperative analgesic requirement
Intraoperative and postoperative side effects | For 24 hours after performing the injection
  These include nausea, vomiting, hypotension, bradycardia, respiratory depression, Hypertension
Time to mobilization out of bed | For 48 hours after performing the procedure
  will be recorded in minutes from skin closure
Post-anesthesia care unit (PACU) length of stay | For 4 hours after surgery
  will be recorded from time between transfer from the operating room to PACU and discharge

CONTACTS AND LOCATIONS:
Overall Officials: Tarek H Ramadan, MD, Principal Investigator — Lecturer of Anesthesia and Surgical Intensive Care; Reem A AbdelRaouf, MD, Study Director — Lecturer of Anesthesia and Surgical Intensive Care
Locations (1):
- Mansoura University Hospitals, Al Mansurah, DK, Egypt

IPD SHARING:
Plan to Share IPD: Undecided